CLINICAL TRIAL: NCT02290106
Title: Effects of Pitavastatin on Insulin Sensitivity and Liver Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Takara Stanley, Assistant Professor of Pediatrics, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014p-002117
Record Dates: First submitted 2014-11-08; First posted 2014-11-13 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Obesity; Fatty Liver, Nonalcoholic
Keywords: obesity; insulin sensitivity; statin (HMG-CoA Reductase Inhibitor); fatty liver
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease; Insulin Resistance; Fatty Liver | interventions — pitavastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pitavastatin (Experimental): pitavastatin 4mg daily by mouth for 6 months
  Interventions: Drug: pitavastatin
- Placebo (Placebo Comparator): Identical placebo 4mg by mouth daily for 6 months
  Interventions: Other: PLACEBO

INTERVENTIONS:
Drug: pitavastatin
  Other Names: Livalo
  Arms: Pitavastatin
Other: PLACEBO
  Arms: Placebo

SUMMARY:
HMG co-A reductase inhibitors, commonly called statins, are an effective treatment for dyslipidemia and atherosclerotic heart disease with proven mortality benefit. While the lipid-lowering effects of statins are well-known, other metabolic effects, including effects on glucose tolerance and ectopic fat distribution, are less completely understood. Recent studies have shown that some statins may increase the risk of diabetes. Further, research has suggested that statins may have some benefit in nonalcoholic fatty liver disease (NAFLD), a condition associated with obesity that includes increased fat in the liver (steatosis) and, in some cases, inflammation and hepatocellular damage (steatohepatitis). Pitavastatin, approved by the United States Food and Drug Administration (FDA) in 2009, is the most recent statin to enter the market. Unlike most statins, pitavastatin is not primarily metabolized through cytochrome P450 (CYP450), and thus has reduced potential for interactions with other medications that are metabolized by CYP450. Previous studies have suggested that pitavastatin may be neutral to glucose homeostasis and may improve hepatic lipid. Neither of these effects has been proven definitively, however, and the current proposal aims to characterize in detail the effects of pitavastatin on glucose homeostasis, hepatic steatosis, and steatohepatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Men age 40-65yo
2. BMI ≥ 27kg/m2 and waist circumference ≥102cm, high probability risk factors for NAFLD
3. At least one of the following indicating insulin resistance: Fasting glucose ≥100mg/dL and <126mg/dL, HOMA-IR >2.0, and/or 2 hour glucose ≥140mg/dL and <200mg/dL following standard glucose tolerance test.
4. 10-year cardiovascular disease risk ≥5% by American Heart Association(AHA)/American College of Cardiology (ACC) Pooled Cohort Equations CV Risk Calculator or LDL ≥ 100mg/dL
5. No use of any statin within 1 year of study entry and not being actively considered for statin therapy by a treating provider.

Exclusion Criteria:

1. Diagnosis of diabetes or use of anti-diabetic medications.
2. Use of erythromycin, rifampin, cyclosporin, colchicine, or gemfibrozil.
3. Use of statin therapy within 1 year prior to study entry as above. Use of any other lipid-modifying therapy (including fish oil, fibrates, niacin, gemfibrozil) within 6 months of study entry.
4. Contraindication to statin therapy.
5. Creatinine > upper limit of normal or known renal disease
6. AST or ALT > 3 times the upper limit of normal
7. hemoglobin < 10g/dL
8. Contraindication to undergoing a magnetic resonance scan.
9. Atherosclerotic cardiovascular disease or low-density lipoprotein cholesterol (LDL-C) ≥ 190mg/dL.
10. Triglyceride ≥500mg/dL

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Grinspoon, MD, Principal Investigator — Massachusetts General Hospital; Takara L Stanley, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Braun LR, Feldpausch MN, Czerwonka N, Weiss J, Branch K, Lee H, Martinez-Salazar EL, Torriani M, Sponseller CA, Grinspoon SK, Stanley TL. Effects of Pitavastatin on Insulin Sensitivity and Liver Fat: A Randomized Clinical Trial. J Clin Endocrinol Metab. 2018 Nov 1;103(11):4176-4186. doi: 10.1210/jc.2018-01446. PMID 30239757

RESULTS

PARTICIPANT FLOW:
Groups:
- Pitavastatin: pitavastatin 4mg daily by mouth for 6 months
  pitavastatin
- Placebo: Identical placebo 4mg by mouth daily for 6 months
  PLACEBO
Period: Overall Study
Arm/Group | Pitavastatin | Placebo
Started | 25 | 25
Completed | 24 | 23
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: (All randomized participants participated in baseline assessments.)
Groups:
- Total: Total of all reporting groups
Arm/Group | Pitavastatin | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (6.5) | 52.9 (7) | 52.8 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 25 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24 | 21 | 45
  Non-white | 1 | 3 | 4
  Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Low density lipoprotein cholesterol (LDL-C, mg/dL) [Mean (Standard Deviation); unit: mg/dL] — Population: Only participants with baseline and final data were used in the calculation of baseline timepoints.
  mg/dL
    number analyzed (Participants) | 24 | 23 | 47
    (all) | 116 (18) | 125 (22) | 120 (20)
Fasting glucose (mg/dL) [Mean (Standard Deviation); unit: mg/dL] — Population: Only participants with baseline and final data were used in the calculation of baseline timepoints.
  mg/dL
    number analyzed (Participants) | 24 | 23 | 47
    (all) | 98 (9) | 97 (9) | 97 (9)
Homeostasis model of insulin resistance (HOMA-IR) [Mean (Standard Deviation); unit: HOMA-IR Score] — Population: Only participants with baseline and final data were used in the calculation of baseline timepoints.
  HOMA-IR Score
    number analyzed (Participants) | 24 | 23 | 47
    (all) | 2.1 (1.9) | 1.6 (1.0) | 1.8 (1.5)
Liver fat content (hepatic fat fraction, %) [Mean (Standard Deviation); unit: %] — This is the percent liver fat content as measured by magnetic resonance spectroscopy technique Population: Only participants with baseline and final data were used in the calculation of baseline timepoints. Five additional participants (1 pitavastatin & 4 placebo) were unable to complete MRI due to inability to fit in the scanner or unanticipated claustrophobia, and 1 scan had unusable data due to technical error.
  %
    number analyzed (Participants) | 23 | 18 | 41
    (all) | 17 (11) | 14 (11) | 16 (11)

OUTCOME MEASURES:

1. Primary Outcome: Insulin-stimulated Glucose Uptake
Description: insulin-stimulated glucose uptake measured by euglycemic hyperinsulinemic clamp
Time Frame: 6 months
Population: All patients with results for baseline and final. In addition to 3 participants who did not finish the study, 2 participants were unable to undergo clamp.
Measure: Mean (Standard Deviation); unit: mg/kg/minute
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 22 | 23
mg/kg/minute | 5.9 (2.1) | 5.9 (1.6)

2. Primary Outcome: Liver Fat
Description: liver fat content as measured by 1H-magnetic resonance spectroscopy
Time Frame: 6 months
Population: All participants with baseline and final data were analyzed. In addition to patients who discontinued from the study, some patients were unable to have MRI scan due to inability to fit in the scanner or unanticipated claustrophobia.
Measure: Mean (Standard Deviation); unit: % liver fat (hepatic fat fraction)
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 21 | 18
% liver fat (hepatic fat fraction) | 17 (11) | 14 (10)

3. Secondary Outcome: Alanine Aminotransferase (ALT)
Description: alanine aminotransferase at the 6 month timepoint
Time Frame: 6 months
Population: all patients with available data at baseline and final
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 24 | 23
U/L | 37 (38) | 27 (17)

4. Secondary Outcome: Aspartate Aminotransferase (AST)
Description: aspartate aminotransferase at 6 month timepoint
Time Frame: 6 months
Population: all patients with available data at baseline and final
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 24 | 23
U/L | 31 (23) | 26 (12)

5. Secondary Outcome: Hepatic Insulin Sensitivity
Description: hepatic insulin sensitivity assessed by glucose infusion rate corrected for fluctuations in serum glucose ("M") during low-dose insulin clamp
Time Frame: 6 months
Population: all patients with available data at baseline and final (note, in addition to 3 patients who discontinued, some patients were unable to undergo clamp procedure)
Measure: Mean (Standard Deviation); unit: mg/kg/minute
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 20 | 22
mg/kg/minute | 1.5 (1.0) | 1.6 (0.7)

6. Secondary Outcome: Hemoglobin A1c (HbA1c)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: % (hemoglobin A1c)
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 24 | 23
% (hemoglobin A1c) | 5.7 (0.5) | 5.7 (0.3)

7. Secondary Outcome: Quantitative Insulin Sensitivity Check Index (QUICKI)
Description: quantitative insulin sensitivity check index (QUICKI) at 6 months. Measure = 1/((log(glucose in mg/dL) + log(insulin in uU/mL))
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: QUICKI index
Arm/Group | Pitavastatin | Placebo
Number analyzed (Participants) | 21 | 23
QUICKI index | 0.16 (0.02) | 0.15 (0.02)

ADVERSE EVENTS:
Time Frame: 6 months (during study period)
Description: Patients were asked at every study visit to recall any adverse events. (Patients were not contacted following study completion.)
Arm/Group | Pitavastatin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/25 | 1/25
Other Adverse Events (participants affected / at risk) | 16/25 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pitavastatin (N=25) | Placebo (N=25)
Chest Pain (General disorders) | 1 (1) | 0 (0) — Acute chest pain with overnight hospitalization; cardiac etiology ruled out with normal cardiac enzymes and other testing
Pancreatic Cancer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pitavastatin (N=25) | Placebo (N=25)
Diarrhea or Loose Stools (Gastrointestinal disorders) | 3 | 7
Any Gastrointestinal Symptoms (Gastrointestinal disorders) | 5 | 8
Any Musculoskeletal Symptoms (Musculoskeletal and connective tissue disorders) | 4 | 6
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 4 | 4
Fatigue (General disorders) | 2 | 5
Headache (Nervous system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT02290106/Prot_SAP_000.pdf